CLINICAL TRIAL: NCT07216521
Title: Optimizing Preoperative Surgical Decision-making for Intraductal Papillary Mucinous Neoplasms: The Role of Intent of Surgery
Brief Title: Intent of Surgery for IPMN
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 25-00989
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Intraductal Papillary Mucinous Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — This study will conduct cyst fluid analysis (CEA, amylase, DNA markers if available).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent surgical resection for IPMN: Pathology reports on patients (18 years old of greater) who underwent surgical resection for IPMN will be accessed for analysis.

SUMMARY:
This multicenter retrospective observational cohort study seeks to:

1. Classify surgical intent in patients with resected Intraductal Papillary Mucinous Neoplasms (IPMN) and quantify the proportion of IPMN-associated cancers diagnosed as overt pancreatic cancer with incidental IPMN association on pathology.
2. Compare clinicopathologic features and outcomes between surveillance-detected and incidentally detected IPMN-derived pancreatic cancers.
3. Revise and redefine risk features limited to patients undergoing surgery for IPMN-related indications, identifying optimal predictors of malignant IPMN (high-grade dysplasia or invasive cancer).

ELIGIBILITY:
Inclusion Criteria:

* All patients (18 years old of greater) who underwent surgical resection for IPMN (including low-, high-grade dysplasia, or invasive carcinoma) between July 1, 2015 and July 1, 2025.

Exclusion Criteria:

* Patients with concomitant pancreatic ductal adenocarcinoma (PDAC)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (18 years old of greater) who underwent surgical resection for IPMN (including low-, high-grade dysplasia, or invasive carcinoma) between July 1, 2015 and July 1, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Grade of IPMN on Final Pathology | Day 0 (Retrospective Analysis)

SECONDARY OUTCOMES:
Recurrence Free Survival | Day 0 (Retrospective Analysis)
  Length of time from surgery for IPMN to recurrence.
Overall Survival | Day 0 (Retrospective Analysis)
  Length of time from surgery to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Sacks, MD MPH PhD, Principal Investigator — NYU Langone Health
Locations (14):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Nanjing University, Nanjing, China
- Heidelberg University, Heidelberg, Germany
- Italy (2):
  - San Raffaele Hospital, Milan
  - Padua University, Padua
- Netherlands (2):
  - University of Amsterdam, Amsterdam
  - University of Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Multicenter collaboration limited by data use agreements between institutions for multicenter data to be used solely for study in question.